CLINICAL TRIAL: NCT05757700
Title: A Phase I Study of T-cell Receptor Alpha Constant (TRAC) Locus Integrated CD19-Targeted 19(T2)28z1xx Chimeric Antigen Receptor (CAR) Modified T Cells in Adult Patients With CD19+ Relapsed or Refractory Large B-Cell Lymphoma
Brief Title: Study of 19(T2)28z1xx TRAC-Chimeric Antigen Receptor (CAR) T Cells in People With B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-401
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: B-Cell Lymphoma; Large B-cell Lymphoma; DLBCL, Nos Genetic Subtypes; High-grade B Cell Lymphoma; Mediastinal Large B-cell Lymphoma
Keywords: B-Cell Lymphoma; Large B-cell Lymphoma; DLBCL; High-grade B cell lymphoma; Mediastinal Large B-cell Lymphoma; TRAC-CAR T cells; Memorial Sloan Kettering Cancer Center; 22-401
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Diffuse Large B-Cell Lymphoma (DLBCL) and large B cell lymphoma (Experimental): Participants have histologically confirmed DLBCL and large B cell lymphoma. Participants will be treated with escalating doses of modified T cells.
  Interventions: Biological: 19(T2)28z1xx TRAC T cell

INTERVENTIONS:
Biological: 19(T2)28z1xx TRAC T cell — Participants will be treated with escalating doses of modified T cells.
  Dose level -1: 3 x 10^6 Dose level 1: 10 x 10^6 Dose level 2: 30 x 10^6 Dose level 3: 100 x 10^6

SUMMARY:
The purpose of this research is to evaluate if study therapy, 19(T2)28z1xx TRAC-chimeric antigen receptor (CAR) T cells, may be an effective treatment for people with relapsed/refractory B-cell lymphoma. Researchers will also evaluate if this study therapy is safe, and to look for the highest dose that causes few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Creatinine ≤1.5 mg/100 ml or creatinine clearance ≥ 45ml/min/m2 , direct bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x upper limit of normal (ULN)
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry.
* Histologically confirmed DLBCL and large B cell lymphoma, including

  * DLBCL, not otherwise specified (NOS), or
  * Transformed DLBCL from follicular lymphoma, or
  * High-grade B cell lymphoma (excluding Burkitt's lymphoma), or
  * Primary mediastinal large B cell lymphoma

AND

* Chemotherapy refractory disease, defined as a failure to achieve at least a partial response or disease progression within 12 months to the last therapy, OR
* Disease progression or recurrence in ≤12 months of prior autologous stem cell transplant (ASCT), OR
* Relapsed disease after 2 or more prior chemoimmunotherapies with at least one containing an anthracycline and CD20 directed therapy

  * Patients need to have radiographically documented disease

Exclusion Criteria:

* ECOG performance status ≥2.
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Active CNS disease
* Impaired cardiac function (LVEF <40%) as assessed by ECHO or MUGA scan.
* Patients with the following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction ≤6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration ≤6 months prior to enrollment
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible.
* Patients with prior allogeneic hematopoietic stem cell transplant are eligible, if more than 3 months from transplant and if patients have no active graft versus host disease (GvHD) and not on systemic immunosuppressive therapy.
* Prior CD19-directed therapy including commercially approved or investigational CD19 CAR T cells or BiTEs is allowed, as long as expression of CD19 is confirmed by flow cytometry or immunohistochemistry.
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection are ineligible.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of the skin.
* Patients with presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, severe brain injuries are ineligible.
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 1 year
  The target toxicity rate for the MTD is

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org